CLINICAL TRIAL: NCT06572696
Title: Ultrasonographic Evaluation of Asymptomatic Shoulder Joint Pathologies in Rheumatoid Arthritis Patients Compared to Healthy Controls: Case-Controlled Study
Brief Title: Ultrasonographic Evaluation of Asymptomatic Shoulder Joint Pathologies in Rheumatoid Arthritis Patients
Acronym: UEASJPRAP
Status: Recruiting | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FSMMD
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Rheumatoid Arthritis; Shoulder Injuries and Disorders
Keywords: Rheumatoid arthritis; shoulder; shoulder impingement syndrome
MeSH Terms: conditions — Arthritis, Rheumatoid; Shoulder Injuries; Disease; Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis Patients: Tuberculum greater cortical surface irregularity, biceps and supraspinatus tendinopathy, supraspinatus and subscapularis dynamic compression and acromiohumeral distance will be evaluated bilaterally by ultrasound.
  Interventions: Diagnostic Test: Shulder Ultrasound
- Healthy individuals: Tuberculum greater cortical surface irregularity, biceps and supraspinatus tendinopathy, supraspinatus and subscapularis dynamic compression and acromiohumeral distance will be evaluated bilaterally by ultrasound.
  Interventions: Diagnostic Test: Shulder Ultrasound

INTERVENTIONS:
Diagnostic Test: Shulder Ultrasound — Ultrasound Shoulder Pathology Rating Scale (USPRS) will be used in the evaluation. While the participants are in a sitting position; A total of 5 variables, including bicipital tendinopathy, supraspinatus tendinopathy, greater tuberculum cortical surface irregularity, supraspinatus dynamic and subscapularis dynamic examination, are evaluated and scored according to the level of pathology; The total USPRS score is obtained by adding the scores of all variables.
  Another parameter evaluated by ultrasonography in this study is the acromiohumeral distance measurement. In AH distance measurement with MSK-US, two measurements will be made with all participants in a neutral resting position and their hands at the top of the circle with the elbow angle of 110 °. In both positions, the probe will be placed longitudinally at the lateral point of the acromion determined by palpation, the distance determined between the acromion and the humeral head will be displayed and measured.

SUMMARY:
Ultrasonographic determination of changes and degree of damage in asymptomatic shoulder joint periarticular structures in RA patients and comparison with healthy controls.

DETAILED DESCRIPTION:
It was designed as a prospective single-blind case-controlled clinical study. Written informed consent was obtained from all study participants who met the study criteria and agreed to participate in the study.

30 RA patients between the ages of 18-75 who had been diagnosed with RA for at least 12 months according to the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) criteria and had no complaint of shoulder pain; Patients will be randomly assigned to the patient group according to the order in which they arrive at the outpatient clinic, regardless of age, gender and disease activation. Exclusion criteria for the study include patients with clinically suspected shoulder pathology, a history of previous shoulder surgery, a history of direct trauma to the shoulder, a history of infectious arthritis, other connective tissue diseases, serious and chronic somatic or psychiatric diseases, any previous fracture in the upper extremities, and patients with limited joint movement.

Healthy volunteers who do not have any complaints or problems regarding the shoulder area will be included in the control group, consisting of a total of 30 participants with similar age, gender and non-RA comorbidities as the RA patient group. Exclusion criteria are the same as the exclusion criteria for the RA patient group.

Demographic data of RA and healthy volunteers such as age, height, weight, body mass index (BMI), gender, marital status, education level, occupation and dominant hand will be recorded. Joint examinations will be performed by an experienced rheumatologist to evaluate the patients' sensitive and swollen joints. The medical history of the patients with RA, including the duration of the disease and the medications they use, and the shoulder joint examination of all participants will be performed by the same physical medicine and rehabilitation specialist doctor blinded to the patient and healthy volunteers. During the examination, joint range of motion (ROM) which include active and passive flexion, extension, abduction, internal and external rotation movements of the shoulder and special tests (Hawkins, Neer, Jobe, Patte, Yergason, Gerber) will be used.

US evaluation of both shoulders of all participants will be performed by the same experienced doctor with more than 5 years of experience in this field, using the MyLab60 brand US machine with a 7-12 MHz superficial probe. The physician performing the evaluation will be blinded to the participants. In order to evaluate intra-rater reliability, measurements will be made twice on 5 patients, 1 day apart.

Ultrasound Shoulder Pathology Rating Scale (USPRS) will be used in the evaluation. USPRS consists of 3 static and 2 dynamic examinations. Static tests; It consists of evaluation of greater tuberculum cortical surface irregularity, biceps and supraspinatus tendinopathy. Dynamic tests are performed to evaluate supraspinatus and subscapularis compression by having the patient abduct and externally rotate, respectively. The USPRS score varies between 0-20 points, while 0 points indicate no pathology, 20 points indicate the highest level of pathology in all variables. While the participants are in a sitting position; A total of 5 variables, including bicipital tendinopathy, supraspinatus tendinopathy, greater tuberculum cortical surface irregularity, supraspinatus dynamic and subscapularis dynamic examination, are evaluated and scored according to the level of pathology; The total USPRS score is obtained by adding the scores of all variables.

Another parameter evaluated by ultrasonography in this study is the acromiohumeral distance (AHM) measurement. One of the most common causes of shoulder pain is subacromial impingement syndrome, and AHM measurement with musculoskeletal ultrasound (MSK-US) is important as it is also a two-dimensional linear measurement of the subacromial area and a marker of rotator cuff diseases. In AH distance measurement with MSK-US, two measurements will be made with all participants in a neutral resting position and their hands at the top of the circle with the elbow angle of 110 °. In both positions, the probe will be placed longitudinally at the lateral point of the acromion determined by palpation, the distance determined between the acromion and the humeral head will be displayed and measured.

ELIGIBILITY:
Inclusion Criteria:

* RA patients between the ages of 18-75 who has been diagnosed with RA for at least 12 months according to the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) criteria and has no complaint of shoulder pain.

Exclusion Criteria:

* Patients with clinically suspected shoulder pathology, a history of previous shoulder surgery, a history of direct trauma to the shoulder, a history of infectious arthritis, other connective tissue diseases, serious and chronic somatic or psychiatric diseases, any fracture in the upper extremities, and patients with limited joint movement.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: RA patients and healthy volunteers(have close demographic data with RA patients)
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2024-09-02 (Estimated); Study Completion 2024-09-02 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Shoulder Pathology Rating Scale | 20 minute
  Ultrasound Shoulder Pathology Rating Scale point

SECONDARY OUTCOMES:
Acromiohumeral Distance | 5 minute
  Acromiohumeral Distance millimetric measurement

CONTACTS AND LOCATIONS:
Overall Officials: Yunus Emre Dogan, MD, Principal Investigator — Istanbul Fatih Sultan Mehmet Training and Research Hospital; Muhsin Doran, MD, Study Chair — Istanbul Liv Hospital; Cigdem Cinar, Assoc Prof, Study Chair — Istanbul Biruni University; Burak Kutuk, MD, Study Chair — Hatay Defne State Hospital
Locations (1):
- Istanbul Physıcal Therapy And Rehabılıtatıon Traınıng And Research Hospıtal, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smolen JS, Aletaha D, Bijlsma JW, Breedveld FC, Boumpas D, Burmester G, Combe B, Cutolo M, de Wit M, Dougados M, Emery P, Gibofsky A, Gomez-Reino JJ, Haraoui B, Kalden J, Keystone EC, Kvien TK, McInnes I, Martin-Mola E, Montecucco C, Schoels M, van der Heijde D; T2T Expert Committee. Treating rheumatoid arthritis to target: recommendations of an international task force. Ann Rheum Dis. 2010 Apr;69(4):631-7. doi: 10.1136/ard.2009.123919. Epub 2010 Mar 9. PMID 20215140
- [Background] Filippucci E, Iagnocco A, Meenagh G, Riente L, Delle Sedie A, Bombardieri S, Valesini G, Grassi W. Ultrasound imaging for the rheumatologist VII. Ultrasound imaging in rheumatoid arthritis. Clin Exp Rheumatol. 2007 Jan-Feb;25(1):5-10. PMID 17417983
- [Background] Filippucci E, Meenagh G, Delle Sedie A, Salaffi F, Riente L, Iagnocco A, Scire CA, Montecucco C, Bombardieri S, Valesini G, Grassi W. Ultrasound imaging for the rheumatologist. XX. Sonographic assessment of hand and wrist joint involvement in rheumatoid arthritis: comparison between two- and three-dimensional ultrasonography. Clin Exp Rheumatol. 2009 Mar-Apr;27(2):197-200. PMID 19473557
- [Background] Abdelzaher MG, Tharwat S, AbdElkhalek A, Abdelsalam A. Ultrasound versus magnetic resonance imaging in the evaluation of shoulder joint pathologies in a cohort of rheumatoid arthritis patients. Int J Rheum Dis. 2019 Dec;22(12):2158-2164. doi: 10.1111/1756-185X.13728. Epub 2019 Oct 31. PMID 31670481